CLINICAL TRIAL: NCT05722353
Title: IBD Disease Course of Infliximab-naïve IBD Patients Treated With Subcutaneous Infliximab CT-P13 Remsima®
Acronym: PRIME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP211343; 2022-A01567-36 (Other: ANSM)
Record Dates: First submitted 2022-08-22; First posted 2023-02-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory bowel disease; Crohn Disease; Colitis; Ulcerative; Infliximab
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Collection of clinical parameters, blood and stools samples (Other): Collection of blood samples and feces specimen at inclusion visit; clinical and biological assessment at each visit.
  Interventions: Other: Biocollection

INTERVENTIONS:
Other: Biocollection — Collection of blood samples and feces specimen at inclusion visit; clinical and biological assessment at each visit.

SUMMARY:
CURRENT STATE OF KNOWLEDGE IN VIEW OF THE RESEARCH About the condition under investigation Inflammatory bowel diseases (IBD), including Crohn's disease and ulcerative colitis, are chronic diseases characterized by relapsing and remitting episodes.

About comparator strategies/procedures Infliximab in its Intravenous (IV) form was the first biotherapy to be approved to treat IBD. Biosimilars of intravenous (IV) infliximab have been shown to be non-inferior to the reference product in patients with IBD, to induce and maintain clinical response

Recently, the subcutaneous (SC) formulation of the infliximab biosimilar CT-P13 (CT-P13 SC) has been shown to be non-inferior on CT-P13 concentration at week 22 to the IV formulation of CT-P13 (CT-P13 IV). These results were based on 66 patients treated with CT-P13 SC, and larger studies are needed to better assess IBD disease course of patients treated with CT-P13 SC in real-life setting.

DETAILED DESCRIPTION:
The study assesses in real-life setting the IBD disease course of infliximab-naïve IBD patients treated with subcutaneous infliximab. This study will look at the clinical and biological outcomes of people who take subcutaneous infliximab.

The study will enroll approximately 120 participants with an indication for iv infliximab.

All participants will receive 1 intravenous infusion on Day 1 and Week 2, followed by 1 SC injection on Week 6 and then 1 SC injection every 2 weeks for up to Week 48.

Switch to subcutaneous infliximab (Remsima® SC) at week 6 will be proposed as part of standard of care.

This multi-center trial will be conducted in hospitals of Assistance Publique - Hôpitaux de Paris (AP-HP). The overall time to participate in this study is 48 weeks. Participants will make approximately 5 visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease or ulcerative colitis (confirmed by clinical evaluation and a combination of endoscopic, histological, radiological, and/or biochemical investigations according to European guidelines)
* Starting infliximab as standard of care (originator or biosimilars)
* with or without concomitant immunosuppressive agent and/or steroids use at infliximab initiation
* Patients agreeing to participate

Exclusion Criteria:

* Patients not eligible to infliximab according to standard of care screening
* Previous exposure to infliximab: originator or biosimilars
* Participation in another interventional study
* No coverage by the French health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Steroids Steroid-free clinical remission defined as Crohn's Disease Activity Index (CDAI) < 150 in patients with CD | week 48
Steroids Steroid-free clinical remission defined as Simple clinical colitis activity index (SCCAI) < 3 in patients with UC | week 48

SECONDARY OUTCOMES:
Clinical response defined as a decrease in CDAI ≥100 from the baseline CDAI score in patients with CD | Week 48
Clinical response defined as a decrease in SCCAI ≥ 3 from the baseline SCCAI score in patients with UC | Week 48
Biological remission | Week 48
  Biological remission is based on CRP level < 5mg/dL
Percentage of patients who switch back to IV infliximab | Week 48
  Percentage of patients who switch back to IV infliximab
clinical relapse-free rates | Week 48
  Relapse will be based on physician global assessment
loss of response rates | Week 48
  loss of response rates at week 48
clinical remission | Week 12
  clinical response and remission
Mean change from baseline in CDAI score in patients with CD | Week 48
Mean change from baseline in SCCAI score in patients with UC | Week 48
Mean change from baseline in CRP | Week 48
Mean change from baseline in fecal calprotectin | Week 48
infliximab through levels | Week 48
Development of anti-infliximab antibodies | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Julien Kirchgesner, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Saint Antoine Hospital Service de Gastroentérologie et Nutrition, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095
- [Background] Hanauer SB, Feagan BG, Lichtenstein GR, Mayer LF, Schreiber S, Colombel JF, Rachmilewitz D, Wolf DC, Olson A, Bao W, Rutgeerts P; ACCENT I Study Group. Maintenance infliximab for Crohn's disease: the ACCENT I randomised trial. Lancet. 2002 May 4;359(9317):1541-9. doi: 10.1016/S0140-6736(02)08512-4. PMID 12047962
- [Background] Ye BD, Pesegova M, Alexeeva O, Osipenko M, Lahat A, Dorofeyev A, Fishman S, Levchenko O, Cheon JH, Scribano ML, Mateescu RB, Lee KM, Eun CS, Lee SJ, Lee SY, Kim H, Schreiber S, Fowler H, Cheung R, Kim YH. Efficacy and safety of biosimilar CT-P13 compared with originator infliximab in patients with active Crohn's disease: an international, randomised, double-blind, phase 3 non-inferiority study. Lancet. 2019 Apr 27;393(10182):1699-1707. doi: 10.1016/S0140-6736(18)32196-2. Epub 2019 Mar 28. PMID 30929895
- [Background] Schreiber S, Ben-Horin S, Leszczyszyn J, Dudkowiak R, Lahat A, Gawdis-Wojnarska B, Pukitis A, Horynski M, Farkas K, Kierkus J, Kowalski M, Lee SJ, Kim SH, Suh JH, Kim MR, Lee SG, Ye BD, Reinisch W. Randomized Controlled Trial: Subcutaneous vs Intravenous Infliximab CT-P13 Maintenance in Inflammatory Bowel Disease. Gastroenterology. 2021 Jun;160(7):2340-2353. doi: 10.1053/j.gastro.2021.02.068. Epub 2021 Mar 5. PMID 33676969